CLINICAL TRIAL: NCT05737641
Title: Ultrasonographic Evaluation of Gastric Content and Volume After Oral Ingestion of Water or Jelly in Volunteers - A Randomised Controlled Non-inferiority Clinical Trial
Brief Title: Gastric Volume After Water or Jelly Ingestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar de Entre o Douro e Vouga (Other)
Responsible Party: Principal Investigator, Paulo Jorge Gomes Correia, Dr. Paulo Correia, Centro Hospitalar de Entre o Douro e Vouga
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CES 48_2022
Record Dates: First submitted 2022-12-23; First posted 2023-02-21 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Fasting; Surgery; Ultrasound Therapy; Complications; Aspiration Pneumonia Due to Regurgitated Food
Keywords: Preoperative Fasting; Elective Surgery; Ultrasound; Gastric Volume; Jelly; Regurgitation; Aspiration pneumonia
MeSH Terms: conditions — Fasting; Gastroesophageal Reflux; Pneumonia, Aspiration

STUDY DESIGN:
Intervention Model Description: RCT crossover study
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- water ingestion (Active Comparator): Ingestion of 102 mL of fresh water
  Interventions: Other: water ingestion
- jelly ingestion (Experimental): ingestion of 100 gr strawberry jelly
  Interventions: Dietary Supplement: jelly ingestion

INTERVENTIONS:
Other: water ingestion — ingestion of water after an 8h-fasting period
  Arms: water ingestion
Dietary Supplement: jelly ingestion — ingestion of jelly after an 8h-fasting period
  Arms: jelly ingestion

SUMMARY:
The aim of this study is to determine whether the fasting duration required for patients after consuming oral jelly is comparable to that after consuming water, prior to elective surgery.

International guidelines for perioperative fasting recommend abstaining from clear fluids for 2 hours to minimize the risk of regurgitation and aspiration pneumonia. However, there are no specific recommendations regarding the perioperative management of jelly consumption.

Current understanding emphasizes the benefits of minimizing preoperative fasting time, including preventing dehydration and metabolic complications like ketoacidosis, as well as potentially enhancing patient satisfaction.

Oral jelly consumption may offer advantages by improving preoperative hydration and providing some nutritional support prior to procedures.

This crossover study will involve 25 adult volunteers. In the first phase, participants will be randomly assigned to either oral intake of water or jelly, followed by the opposite intervention in the second phase. Gastric content and volume will be assessed using gastric ultrasound.

DETAILED DESCRIPTION:
Prolonged preoperative fasting is associated with unfavorable outcomes, inducing a catabolic state that may lead to metabolic disturbances such as ketoacidosis, insulin resistance, dehydration, and increased postoperative complications such as surgical site infection and delayed bowel function. To minimize fasting time, current guidelines from the American Society of Anesthesiology advise clear fluid intake (water, tea, coffee, pulp-free fruit juices, carbohydrate-rich beverages) up to 2 hours prior to elective procedures involving general anesthesia, regional anesthesia, or procedural sedation and analgesia. Solids fasting should extend to 6 to 8 hours, depending on the type of foods.

Jelly is a solid food, mostly composed of water. Among its other components, proteins, responsible for its solidification, and sugars stand out. Thus, it may be a form of oral hydration, associated with some nutritional value, but the appropriate preoperative fasting time is not explicitly stated in the guidelines.

An important cause of mortality and morbidity associated with tracheal intubation is the aspiration of gastric contents. It is important to ensure that restricting preoperative fasting time does not compromise patient safety, thereby increasing this risk. While carbohydrate-rich beverages are not associated with delays in gastric emptying, the same cannot be said for protein-containing liquids.

Gastric ultrasound is a non-invasive, bedside-available, and reliable method for quantitative and qualitative assessment of stomach contents. Although the minimum volume of gastric contents associated with increased risk of aspiration is not known, some studies demonstrate that volumes up to 1.5 mL/kg of clear fluids, in the absence of solid contents, are normal, commonly seen in fasting adults, and are not associated with an increased risk of pulmonary aspiration.

The aim of our study is to demonstrate that jelly ingestion, compared to water, is not associated with larger cross-sectional area of the gastric antrum, behaving similarly to clear fluids.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers working in the hospital Centro Hospitalar de Entre o Douro e Vouga (CHEDV)

Exclusion Criteria:

* morbid obesity
* pregnancy
* alcohol abuse
* diseases or drugs that can prolong or accelerate gastric emptying such as gastric or esophageal surgery, diabetes mellitus, prokinetic or opioid use, hypothyroidism
* intolerance to any of the components of jelly

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
gastric antral cross-sectional area | 2 hours after intervention
  antral cross-sectional area measured by ultrasound in right lateral decubitus position (non-inferiority test)

SECONDARY OUTCOMES:
gastric volume | 2 hours after intervention
  gastric volume calculated by the formula of Perlas et al
gastric volume greater than 1.5 mL/Kg | 2 hours after intervention
  number of participants with gastric volume greater than 1.5 mL/kg
Qualitative gastric evaluation | 2 hours after intervention
  Empty, fluid or solid
hunger and thirst | 2 hours after intervention
  hunger and thirst on a visual analogue scale from 0 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar de Entre Douro e Vouga (CHEDV), Santa Maria da Feira, Aveiro District, Portugal

IPD SHARING:
Plan to Share IPD: No